CLINICAL TRIAL: NCT01855009
Title: A Comparative Effectiveness Research Study Comparing Changes in Body Composition and Parent Ratings of Quality of Life in 5-19 Year Olds as a Function of Participation in One of Four Versions of the Good NEWS 4 Kids Program (GN4K)
Brief Title: Study of Parental Ratings of Quality of Life and Body Composition in 5-19 Year Olds While Participating in the Good NEWS 4 Kids Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Health Technologies, Inc. (Network)
Collaborators: MannaRelief Ministries (Unknown)
Responsible Party: Principal Investigator, Gilbert R Kaats, Dr. Gilbert R. Kaats, PhD, Integrative Health Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 066
Record Dates: First submitted 2013-05-08; First posted 2013-05-16 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Quality of Life; Body Mass Index
Keywords: Quality of Life; Body Weight and Measures; Malnutrition; Adolescent Nutrition Sciences; Sleep Initiation and Maintenance Disorder; Motor Activity; Drinking
MeSH Terms: conditions — Body Weight; Malnutrition; Motor Activity | interventions — Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MannaBears (Active Comparator): Subjects will take 4 MannaBears daily
  Interventions: Dietary Supplement: MannaBears
- MannaBears, AlgaeCal Calcium, Vitamin D3 (Active Comparator): Subjects will take 4 MannaBears daily and 3 Calcium/Vit D capsules (2 with breakfast and 1 with dinner or vice-versa) daily
  Interventions: Dietary Supplement: MannaBears; Dietary Supplement: AlgaeCal Calcium; Dietary Supplement: Vitamin D3
- MannaBears, Calcium Carbonate, Vitamin D3 (Active Comparator): Subjects will take 4 MannaBears daily and 3 Calcium/Vit D capsules (2 with breakfast and 1 with dinner or vice-versa) daily
  Interventions: Dietary Supplement: MannaBears; Dietary Supplement: Calcium carbonate; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: MannaBears — Subjects will be administered 4 MannaBears daily
Dietary Supplement: AlgaeCal Calcium — Subjects will be administered 750 mg AlgaeCal Calcium
  Arms: MannaBears, AlgaeCal Calcium, Vitamin D3
Dietary Supplement: Calcium carbonate — Subjects will be administered 1000 mg calcium carbonate
  Arms: MannaBears, Calcium Carbonate, Vitamin D3
Dietary Supplement: Vitamin D3 — Subjects will be administered 800 IU vitamin D3
  Arms: MannaBears, AlgaeCal Calcium, Vitamin D3; MannaBears, Calcium Carbonate, Vitamin D3

SUMMARY:
This study will compare changes in body composition (lean mass, fat, and bone)and parent ratings of quality of life in 5-19 Year Olds as a function of participation in one of four versions of the Good NEWS 4 Kids Program (GN4K).

DETAILED DESCRIPTION:
Purpose: The objectives of this study are to:

1. Compare the relative efficacy of four variations of the GN4K program in facilitating positive changes in body composition and parental ratings of quality of life.
2. Compare parental ratings of children's behavior to DXA-measured changes in body composition;
3. Compare measurements of scale weight, height, waist/hip ratios and BMI with DXA-measured changes in body composition;
4. Develop a logarithm formula with the use of anthropometric measurements and parental ratings to predict body composition changes

ELIGIBILITY:
Inclusion Criteria:

* Must ensure with medical provider that there are not medical conditions that would preclude participation
* Must be between the ages of 5 and 19

Exclusion Criteria:

* males and females below the age of 5 and above the age of 19
* pregnant or breast feeding

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in parental ratings of participating child's quality of life | 0 and 90 days
  Parent(s) will complete questionnaires on a monthly basis to assess the improvements made or improvements that have been made in various areas of their child's behavior and activities. Change from baseline to end of study will be reported.

SECONDARY OUTCOMES:
Changes in body composition as a measurement of Dual Energy Absorptiometry | 0 and 90 days
  Body composition (fat, fat-free mass, and bone mineral density) as measured by Dual Energy Absorptiometry (DXA)
Changes in hip to waist ratios | 0 and 90 days
  Parent(s) will be provided with a tape measure with which they will measure their child's hip and waist.
Changes in blood pressure | 0 and 90 days
  Blood pressure will be measured at the time the DXA measurement is completed.
Changes in gender and age adjusted BMI | 0 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert R Kaats, PhD FACN, Principal Investigator — Integrative Health Technologies, Inc.; Harry G Preuss, MD MACN, Study Chair — Georgetown University Medical Center, Dept of Biochemistry, Medicine and Pathology
Locations (1):
- Integrative Health Technologies, San Antonio, Texas, United States